CLINICAL TRIAL: NCT03800732
Title: The Influence of Nocturnal Food Intake in Eating Behavior of Night Workers: Randomized Cross-over Study.
Brief Title: The Influence of Nocturnal Food Intake in Eating Behavior of Night Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Cibele Aparecida Crispim, Principal investigator, Federal University of Uberlandia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 86382218.6.0000.5152
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Shift Work Type Circadian Rhythm Sleep Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Night workers. (Experimental): Night workers of the military police of Minas Gerais, Uberlândia, who will participate in the three interventions of the study.
  Interventions: Other: With Meal during night work; Other: Without Meal during night work; Other: Sleep night

INTERVENTIONS:
Other: With Meal during night work — Two nights of work with a meal during the shift and after will go to the laboratory the morning for eating a test meal ad libitum, which will consist of foods of various compositions and food groups. Preprandial metabolic assessments will be conducted (ghrelin, GLP-1 - glucagon-like peptide 1, PYY-peptide YY). The following postprandial evaluations will be carried out and in the 24 hours following the experiment: food choices (record of all foods) and food perceptions (hunger, appetite, satiety and eating).
Other: Without Meal during night work — Two nights of work without a meal during the shift and after will go to the laboratory the morning for eating a test meal ad libitum, which will consist of foods of various compositions and food groups. Preprandial metabolic assessments will be conducted (ghrelin, GLP-1 - glucagon-like peptide 1, PYY-peptide YY). The following postprandial evaluations will be carried out and in the 24 hours following the experiment: food choices (record of all foods) and food perceptions (hunger, appetite, satiety and eating).
Other: Sleep night — Two sleep nights and after will go to the laboratory the morning for eating a test meal ad libitum, which will consist of foods of various compositions and food groups. Preprandial metabolic assessments will be conducted (ghrelin, GLP-1 - glucagon-like peptide 1, PYY-peptide YY). The following postprandial evaluations will be carried out and in the 24 hours following the experiment: food choices (record of all foods) and food perceptions (hunger, appetite, satiety and eating).

SUMMARY:
This study aimed to verify the influence of night work and food intake during the night shift on the eating behavior of fixed night workers the next day.

DETAILED DESCRIPTION:
Night work causes restriction of sleep time and circadian misalignment and, therefore, have been associated with nutritional and metabolic impairments. The objective of the present study is to verify the influence of night work and food intake in this period on the behavior of the following day. The workers selected by criteria and inclusion and exclusion will be evaluated at the baseline: anthropometric parameters, food consumption and perception, duration of food consumption, sleep habits and chronobiological pattern (sleep monitoring by actigraphy, chronotype, social jet lag), parameters biochemical (blood count, lipidogram, C-reactive protein, cortisol, glucose, insulin).Subsequently, 30 workers will integrate a randomized and controlled crossover clinical study with three randomly established interventions: (1) two nights of work without meals during the shift; (2) two nights of work with a meal during the shift; (3) two nights sleep. Participants will go to the laboratory the morning after the second night of each condition to offer a test meal ad libitum, which will consist of foods of various compositions and food groups. Preprandial metabolic assessments will be conducted (ghrelin, GLP-1 - glucagon-like peptide 1, PYY-peptide YY). The following postprandial evaluations will be carried out and in the 24 hours following the experiment: food choices (record of all foods) and food perceptions (hunger, appetite, satiety and eating). It is expected to determine how nocturnal versus nocturnal work, and nocturnal fasting versus nocturnal fasting affect the next day's food choices.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study and sign the Informed Consent Form (EHIC).
* No significant changes in body mass in the last 6 months.
* With stable food and sleep routine in the last two months.

Exclusion Criteria:

* Failure to provide the information or material necessary for the development of the study.
* Report of chronic non-communicable diseases.
* Report of diagnosed and untreated psychiatric disorders.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Preprandial metabolic | 6 months
  Ghrelin, GLP-1 - glucagon-like peptide 1, PYY-peptide YY
Change of food perceptions | 6 months
  To evaluate appetite, satiety and postprandial satisfaction, a visual analogue scale was applied before and after consumption of the proposed meal, with the questions, "How much hunger did you have before the meal?"; "After the meal, how did you feel?"; "How much did you like the meal?", Signaling all responses on a 0 to 10 cm scale.

SECONDARY OUTCOMES:
Food behavior | 6 months
  Record of food consumption of the meals / snacks held following the test meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Cibele Aparecida Crispim, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Teixeira BS, Silva CM, Silva ATF, Santos LLD, de Paiva Maia YC, Pedrazzoli M, Wright KP Jr, Crispim CA. Influence of fasting during the night shift on next day eating behavior, hunger, and glucose and insulin levels: a randomized, three-condition, crossover trial. Eur J Nutr. 2023 Apr;62(3):1281-1293. doi: 10.1007/s00394-022-03069-6. Epub 2022 Dec 17. PMID 36526739